CLINICAL TRIAL: NCT02528370
Title: Evaluation the Effectiveness of a Telemonitoring Program in a Cohort of COPD Patient With Frequent Readmissions
Acronym: telEPOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Cristobal Esteban (Other Government)
Collaborators: Osakidetza (Other)
Responsible Party: Sponsor-Investigator, Dr. Cristobal Esteban, MD, Hospital Galdakao-Usansolo
Organization: Hospital Galdakao-Usansolo (Other Government)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PI013/02352
Record Dates: First submitted 2015-08-17; First posted 2015-08-19 (Estimated); Results first posted 2021-02-16 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: COPD
Keywords: COPD exacerbation; Telemedicine; Intervention Studies; Patient Readmission
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Only data entry people and biostatisticians were masking
Oversight: Data Monitoring Committee: No

ARMS (2):
- telEPOC (Experimental): The program consisted of: 1) Educational program about COPD. This educational program was carried-out by a respiratory nurse in two 30-minute speeches to the patient and career, once at their inclusion in the program and again 1 year later. 2) Training in using the device (smart phone) that supported the telemonitoring. 3) Daily phone calls to make self-confident the patient during the first week. Afterwards the phone calls were established according to the capacity of the patient to manage on their own.
  Interventions: Device: telEPOC
- No telEPOC / Usual Care (No Intervention): The control group follows the usual care protocol in our health system. That includes periodic control by their primary and respiratory specialist. They receive non-structured information/education about COPD and follow a programmed control agenda depending on the severity of the disease every 4-6 months.
  Generally speaking the differences between the two cohorts were the educational structured program and the telemonitoring control.

INTERVENTIONS:
Device: telEPOC — The program consisted of: 1) Educational program about COPD. This educational program was carried-out by a respiratory nurse in two 30-minute speeches to the patient and career, once at their inclusion in the program and again 1 year later. 2) Training in using the device (smart phone) that supported the telemonitoring. 3) Daily phone calls to make self-confident the patient during the first week. Afterwards the phone calls were established according to the capacity of the patient to manage on their own.
  Arms: telEPOC

SUMMARY:
Observational non-randomized study with an intervention cohort from Hospital Galdakao-Usansolo with 119 patients and a control cohort from Hospital Cruces with 78 patients. The inclusion criteria were: being hospital admitted at least twice in the previous year or at least three times in the 2 previous years. The cohorts were follow-up for 2 years. Several clinical measurements like pulmonary function, exercise capacity, health related quality of life, limitation in daily life activities and anxiety and depression were recorded in both cohorts. Telemonitoring and an organized education program were only and exclusively applied in the intervention cohort.

DETAILED DESCRIPTION:
During July 2010 and July 2013 COPD patients from two health-administrative areas (integrated sanitary organization -ISO-) in Bizkaia were recruited. Each of these two areas is supported by 1 hospital. Hospital Galdakao-Usansolo hospital (ISO-Barrualde), which is in charge of the health of 350000 inhabitants and in the second, hospital Cruces (OSI-Ezkerraldea Cruces) with 350000 inhabitants. The cohort from Galdakao was the intervention cohort while the cohort from Cruces was the control cohort. Both cohorts were followed-up for two years.

Participants The inclusion criteria established were: having a COPD (COPD was confirmed if the post-bronchodilator forced expiratory volume in one second (FEV1) divided by the forced vital capacity (FVC) was less than 0.7 (FEV1/FVC<70%) and having been admitted at least twice in the previous year or three times in the two previous years for a COPD exacerbation (eCOPD). Exclusion criteria were another significant respiratory disease, an active neoplasm, a terminal clinical situation, inability to carry out any of the measurements of the project, or unwillingness to take part in the study.

With these requirements, patients were chosen from the database of the hospital. The potential candidates and their career were informed about the program in a general informative meeting, or individually during an admission, and invited to participate. If the patient wanted to take part in the program they signed the informed consent form.

Usual clinical care At the time of this study COPD patients had no take part in any specific clinical control program in the public health system. Patients were being controlled following a schedule by their primary doctor and respiratory specialist. The frequency of the control depended on the severity of the disease. In case of eCOPD they had to schedule a visit to their primary doctor.

Intervention The patients had to present a stable COPD, at least for six weeks before enrollment. All the participants had a previous spirometry but COPD diagnosis was confirmed at the moment of inclusion in the program.

The program consisted of: 1) Educational program about COPD (general information about what COPD is, general treatment of the disease focusing on tobacco and inhaled medication, life healthy habits and alarm signs related to eCOPD). This educational program was carried-out by a respiratory nurse in two 30-minute speeches to the patient and career, once at their inclusion in the program and again 1 year later. 2) Training in using the device (smart phone) that supported the telemonitoring. 3) Daily phone calls to make self-confident the patient during the first week. Afterwards the phone calls were established according to the capacity of the patient to manage on their own.

Generally speaking during the two years of the program in every phone call patients were given some advice on daily healthy habits, specially physical activity.

Written information about how the program ran and how to use the smart phone as well as a contact phone number was provided to every patient and career.

No home visits were part of the program. No self-management plans of exacerbation were included in the program.

The implementation of this program was previously explained to all the primary doctors in two general meetings.

The program was supported by a specialized respiratory nurse, working in the hospital Galdakao-Usansolo as a full timer and two part-time respiratory physicians working on the program from Monday to Friday. During the evening and at the weekends a centralized call-center (non specialized respiratory nurses) was in charge of the program.

The device was a smart phone with a specific software for the program, including some measurements of physiological variables such as temperature, breath rate, oxygen saturation, heart rate and steps/day) and a clinical questionnaire (characteristics of cough and sputum, level of dyspnea and general clinical health status).

Patients included in the program (telEPOC program) had to send information about their clinical situation on a daily basis. This daily information was sent by a secure internet connection to protect server and transfer to the respiratory service, where a nurse analyzed the whole information of every patient. Every patient had a tailored-made baseline level of these measurements established in a stable clinical situation at the moment of inclusion in the program. This baseline was the reference for the daily measurements. Once the patient´s measurements were received, were automatically ordered in three colored levels (traffic lights) depending of the deviation of the measurement with respect the baseline measurement (alarm). The alarm three levels was established by consensus of the research team depending on the different combination of measurement daily sent by the patients. Once the patient measurements were received, there were several possible actions. If all the data were normal with respect to the personalized threshold previously established, not a single action was done. If the established threshold was surpassed, an alarm was activated and an protocol action plan was started up. The first step was a phone call to the patient or the career. This phone call was used to confirm the alarm and its level of priority and try to solve it as long as it was possible. If this action was not considered useful or did not solve the alarm the nurse had two options, depending on the severity of the alarm, wait for the daily evaluation of the patient bi respiratory physicians (ward daily rounds) or contact one of the respiratory physicians. At this point it was the respiratory physician who determined if the patient should be sent to his primary doctor or be evaluated by a respiratory specialist or sent to the hospital emergency department.

If a patient had to be evaluated by a doctor at the primary level or at a specialized level, the nurse of the program previously contact the doctor to arrange an appointment. An alert system warned the monitoring team if daily measurements had not been submitted.

Primary outcome: The primary outcome of the program was to diminish the rate of hospitalizations for eCOPD. We defined an exacerbation as a sustained worsening of the participant's COPD symptoms from their usual stable state that was beyond normal day-to-day variations, and with a severity level that need hospital admission to be solved.

Control cohort. The control group follows the usual care protocol in our health system. That includes periodic control by their primary and respiratory specialist. They receive non-structured information/education about COPD and follow a programmed control agenda depending on the severity of the disease every 4-6 months. Generally speaking the differences between the two cohorts were the educational structured program and the telemonitoring control.

Baseline assessment The study protocol performed in the intervention and in the control cohort included several measurements before being included in the program and every year during the follow-up.

Sociodemographic variables and smoking habits were recorded. The level of dyspnea was established using modified Medical Research Council score [10]. Comorbidities were determined by reviewing patients' medical records for their clinical histories and Charlson Comorbidity Index calculates. Health related quality of life (HRQoL) was assessed using the Spanish validated version of Saint George's Respiratory Questionnaire (SGRQ) and the COPD Assessment Test (CAT). London Chest Activity of Daily Living scale questionnaire (LCADL). Anxiety and Depression were measured by Hospital Anxiety and Depression (HAD) scale .

Complete pulmonary function tests included forced spirometry, bronchodilator test, body plethysmography, carbon monoxide diffusing capacity, respiratory muscle strength. Theoretical values were those established by the European Community for Steel and Coal.

Two 6-minute walking tests were performed according to American Thoracic Society (ATS) guidelines.

The intervention group daily used a pedometer.

Follow-up In the control cohort every year during the follow-up period, survivors were interviewed and underwent the previously described measurements.

No others interventions were performed related to this study, and the research team did not take part in patients' routine treatment or the treatment of exacerbations. In every visit, reviewing medical reports and examining the hospital database hospitalizations were determined.

Data collection Data about hospitalizations and emergency department admission were collected in real time because the patients were trained to notify these circumstances and the daily follow-up permitted to know the situation of every patient in every moment. Moreover if a patient did not send the daily data the system generated an alarm resulting in a phone call from the nurse to know the reason why the information had not been sent. Besides, in every patient a review of hospital and emergency department admission was carried out at the end of every year.

The questionnaires and pulmonary function test and exercise capacity were performed every year.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria established were: having a COPD (COPD was confirmed if the post-bronchodilator forced expiratory volume in one second (FEV1) divided by the forced vital capacity was less than 0.7 (FEV1/FVC<70%) and having been admitted at least twice in the previous year or three times in the two previous years for a COPD exacerbation (eCOPD).

Exclusion Criteria:

* Exclusion criteria were another significant respiratory disease, an active neoplasm, a terminal clinical situation, inability to carry out any of the measurements of the project, or unwillingness to take part in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2010-05; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cristobal Esteban, MD, Principal Investigator — Staff member

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pinnock H, Hanley J, McCloughan L, Todd A, Krishan A, Lewis S, Stoddart A, van der Pol M, MacNee W, Sheikh A, Pagliari C, McKinstry B. Effectiveness of telemonitoring integrated into existing clinical services on hospital admission for exacerbation of chronic obstructive pulmonary disease: researcher blind, multicentre, randomised controlled trial. BMJ. 2013 Oct 17;347:f6070. doi: 10.1136/bmj.f6070. PMID 24136634
- [Background] Bolton CE, Waters CS, Peirce S, Elwyn G; EPSRC and MRC Grand Challenge Team. Insufficient evidence of benefit: a systematic review of home telemonitoring for COPD. J Eval Clin Pract. 2011 Dec;17(6):1216-22. doi: 10.1111/j.1365-2753.2010.01536.x. Epub 2010 Sep 16. PMID 20846317
- [Background] McLean S, Nurmatov U, Liu JL, Pagliari C, Car J, Sheikh A. Telehealthcare for chronic obstructive pulmonary disease: Cochrane Review and meta-analysis. Br J Gen Pract. 2012 Nov;62(604):e739-49. doi: 10.3399/bjgp12X658269. PMID 23211177
- [Background] McLean S, Sheikh A, Cresswell K, Nurmatov U, Mukherjee M, Hemmi A, Pagliari C. The impact of telehealthcare on the quality and safety of care: a systematic overview. PLoS One. 2013 Aug 19;8(8):e71238. doi: 10.1371/journal.pone.0071238. eCollection 2013. PMID 23977001
- [Derived] Esteban C, Moraza J, Iriberri M, Aguirre U, Goiria B, Quintana JM, Aburto M, Capelastegui A. Outcomes of a telemonitoring-based program (telEPOC) in frequently hospitalized COPD patients. Int J Chron Obstruct Pulmon Dis. 2016 Nov 24;11:2919-2930. doi: 10.2147/COPD.S115350. eCollection 2016. PMID 27920519

RESULTS

PARTICIPANT FLOW:
Groups:
- telEPOC: The program consisted of: 1) Educational program about chronic obstructive pulmonary disease (COPD). This educational program was carried-out by a respiratory nurse in two 30-minute speeches to the patient and career, once at their inclusion in the program and again 1 year later. 2) Training in using the device (smart phone) that supported the telemonitoring. 3) Daily phone calls to make self-confident the patient during the first week. Afterwards the phone calls were established according to the capacity of the patient to manage on their own.
Period: Overall Study
Arm/Group | telEPOC | No telEPOC / Usual Care
Started | 119 | 78
Completed | 102 | 77
Not Completed | 17 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | telEPOC | No telEPOC / Usual Care | Total
Number analyzed (Participants) | 119 | 78 | 197
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.34 (9.36) | 70.1 (7.5) | 70.83 (8.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 10 | 26
  Male | 103 | 68 | 171
Region of Enrollment [Count of Participants; unit: Participants]
  Spain | 119 | 78 | 197
Body mass, airflow obstruction, dyspnea, and exercise capacity (BODE) index [Mean (Standard Deviation); unit: units on a scale] — Total possible values: 0-10 points. Do higher values in each part: worse outcome. All subscales must be summed to calculate the total score.
  * Body mass index:
    0 points:>21
    1 point:≤ 21
  * Degree of airflow obstruction (FEV1% of predicted):
    0 points:≥ 65
    1. point:50-64
    2. points:36-49
    3. points:≤35
  * Dyspnea (mMRC; modified Medical Research Council):
    0 points:0-1
    1. point:2
    2. points:3
    3. points:4
  * Exercise capacity (6MWD; 6-minute walk distance (m)):
    0 points:≥ 350
    1. point:250-349
    2. points:150-249
    3. points:≤149
  Abbreviation: FEV1: forced expiratory volume in one second.
  units on a scale | 4.3 (2.5) | 3.9 (2.2) | 4.1 (2.4)

OUTCOME MEASURES:

1. Primary Outcome: Number of Hospitalizations for COPD Exacerbation (eCOPD)
Description: The primary outcome of the program was to diminish the rate of hospitalizations for eCOPD. We defined an exacerbation as a sustained worsening of the participant's COPD symptoms from their usual stable state that was beyond normal day-to-day variations, and with a severity level that need hospital admission to be solved.
Time Frame: two years
Measure: Mean (95% Confidence Interval); unit: number of hospital admissions
Arm/Group | telEPOC | No telEPOC / Usual Care
Number analyzed (Participants) | 119 | 78
number of hospital admissions | 1.1 [0.7 to 1.5] | 2.8 [2.2 to 3.4]

ADVERSE EVENTS:
Arm/Group | telEPOC | No telEPOC / Usual Care
All-Cause Mortality (participants affected / at risk) | 13/119 | 22/78
Serious Adverse Events (participants affected / at risk) | 2/119 | 0/78
Other Adverse Events (participants affected / at risk) | 0/119 | 0/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | telEPOC (N=119) | No telEPOC / Usual Care (N=78)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0

LIMITATIONS AND CAVEATS:
Our results could probably not be translated to other health systems. We will not be able establish which parts of the results are related to the every part of the program. The level of education of patients may play a role in the results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes